CLINICAL TRIAL: NCT04487002
Title: Outcome After Surgical Treatment of Gastrointestinal Stromal Tumors in the Second Part of Duodenum: Is Localized Resection Appropriate?
Brief Title: Outcome After Surgical Resection of Gastrointestinal Stromal Tumors (GIST) in the Second Part of Duodenum
Acronym: GIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hani Alhadad, assistant professor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 441/11
Record Dates: First submitted 2020-07-18; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Stromal Tumor of Duodenum
Keywords: Gastrointestinal stromal tumor of duodenum; localized resection; survival
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group A (Experimental): underwent localized resection
  Interventions: Procedure: surgical resection

INTERVENTIONS:
Procedure: surgical resection
  Other Names: localized resection or pancreaticoduodenectomy

SUMMARY:
it is hypothesized that long term outcomes of localized resection of GIST tumors located in the second part of the duodenum are comparable to those of the traditional treatment by radical resection of the head o pancreas and the entire duodenum

DETAILED DESCRIPTION:
the Medical records of patient with second part duodenal GIST were reviewed retrospectively for symptoms, clinical examination, preoperative workup including standard imaging by multi-slice computed tomography (CT) of abdomen and pelvis with oral and intravenous contrast. Endoscopic ultrasound was routinely perfumed to assess the depth of tumor invasion (T-stage) and to obtain a tissue sample by fine needle aspiration cytology (FNAC). Definitive diagnosis was based on CT images and post-operative pathology report.

Patients were subjected to curative localized resection with free margins by frozen section examination or pancreaticoduodenectomy (PD) if the tumor was invading the major duodenal papilla.

Localized duodenal resection was performed by one of two techniques: The first one was excision of part of the wall (wedge resection). Reconstruction was performed either by primary closure without tension, provided that adequate lumen is preserved, or by side to side roux-en-Y duodenojejunostomy (DJ) if there was tension on the edges of the duodenal defect. The second technique was employed in case of larger size tumors and entailed excision of D2 (segmental duodenectomy) to be followed by anastomosis (side to side roux-en-Y DJ or end-to-end DJ). Great care to avoid tumor rupture was emphasized in all operations. Standard lymph node dissection was not performed.

Pathologic data (tumor location, size, margins, and mitoses per 50 high-power fields [HPF]) and immunohistochemical analysis were collected and tumors classified into very low, low, moderate and high risk based on Miettinen classification that also incorporates tumor size.

All patients (those who underwent localized resection with safety margin and those who underwent PD) were followed up and re-evaluated at one, three, six and twelve months then once per year for a total follow-up period of 3 years. Contrast-enhanced multi-slice CT abdomen/pelvis was performed after 6 months then yearly for detection of recurrence.

Using PASS program version 20, the minimum sample size required was 45 patients with duodenal GIST using 3% local recurrence rate and 5% error at 5% level of significance and 80% power. Data were analyzed using IBM-SPSS software package version 20. Qualitative variables were summarized using numbers and percent. Quantitative variables were summarized using mean and standard deviation (SD) as data was normally distributed by kolmogrov-smirnov test. Survival analysis was done using life tables, log-rank test and Kaplan Meier's curve. All statistical analysis was conducted at 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* patients with second part duodenal GIST

Exclusion Criteria:

* metastatic, irresectible and unfitness for surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
survival | 3 years
  Survival was calculated from the date of surgery to the time of death
recurrence rate | 3 years
  . Contrast-enhanced multi-slice CT abdomen/pelvis was performed after 6 months then yearly for detection of recurrence

SECONDARY OUTCOMES:
post-operative complications | one month
  leak, wound infection, chest infection

CONTACTS AND LOCATIONS:
Overall Officials: Wael N Abdelsalam, doctor, Study Director — dean of faculty
Locations (1):
- Faculty of Medicine, Alexandria, Egypt